CLINICAL TRIAL: NCT06502041
Title: A Randomized Clinical Trial Comparing MARPE Effect With/Without MOP in Management of Skeletal Transverse Deficiency in Non-growing Patients
Brief Title: MARPE Effect With/Without MOP in Non-growing Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Motaz Elshehaby, principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A05020822
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Maxillary Transverse Deficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of either patient or clinician is not possible. However, blinding was ensured during analyzing the data. All digital models and x-rays were coded and shuffled before they were evaluated and measured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MARPE with MOP (Experimental)
  Interventions: Procedure: MARPE with MOP
- MARPE without MOP (Active Comparator)
  Interventions: Procedure: MARPE without MOP

INTERVENTIONS:
Procedure: MARPE with MOP — mini-screw assisted rapid palatal expansion with micro-osteoperforation
  Arms: MARPE with MOP
Procedure: MARPE without MOP — mini-screw assisted rapid palatal expansion without micro-osteoperforation
  Arms: MARPE without MOP

SUMMARY:
This study compares the effect of MARPE (mini-implant assisted rapid palatal expansion) versus MARPE+ MOP (Micro-osteo-perforation) on nasal airway and maxillary transverse deficiency in non-growing patients.

DETAILED DESCRIPTION:
All participants with skeletal transverse deficiency with unilateral or bilateral cross-bite aging 20-25 years were treated by expansion of maxillary arch as a first phase of treatment with one expander screw which was anchored to mini-implants placed in the palatal region (Mini-implant assissted rapid palatal expansion; MARPE). The patient's bone support in the anterior area of the palate was examined on CBCT. Micro-osteoperforation (MOP) was done along of medial palatine raphe in the intervention group. Control-group is the same of the intervention group but without micro-osteo-perforations.

ELIGIBILITY:
Inclusion Criteria:

1. The age ranges from 20-25 years.
2. Post pubertal adolescent
3. Skeletal transverse deficiency with unilateral or bilateral cross-bite
4. Extraction is not indicated in the lower arch.
5. Upper permanent dentition is erupted up to the second molars.
6. Average facial vertical growth pattern.
7. Space deficiency in the upper arch is less than 8 mm

Exclusion Criteria:

1. Diseases and medications those are likely to affect bone biology.
2. Evidence of root resorption.
3. Poor oral hygiene.
4. Previous orthodontic treatment.
5. Evidence of bone loss.
6. Active periodontal disease.
7. Craniofacial congenital anomalies, such as cleft lip and palate.

7. Pregnant females. 8. Presence of oral habits.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Number of days till diastema appearance | about 1 month
  (days)
Amount of skeletal expansion | about 1 month
  (mm)
Pain experience during activation of expander by visual analogue scale ( VAS) | about 1 months
  VAS: 0 ( no pain), 10 (unbearable pain)
Skeletal, Dental & Nasal readings | measured before treatment and after 6 month of treatment
  from CBCT and scanned models measured in degrees & mm
Stability of correction of transverse deficiency | about 6 months
  by measuring the same CBCT transverse reading and by superimposition of the scaneed models at the end of the research

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Adakhlia, Egypt

IPD SHARING:
Plan to Share IPD: No
the published results

REFERENCES:
- [Derived] Elshehaby M, Albelasy NF, Elbialy MA, Hafez AM, Abdelnaby YL. Evaluation of pain intensity and airway changes in non-growing patients treated by MARPE with and without micro-osteoperforation: a randomized clinical trial. BMC Oral Health. 2024 Nov 20;24(1):1411. doi: 10.1186/s12903-024-05196-4. PMID 39563319